CLINICAL TRIAL: NCT05930145
Title: A Randomized Study Comparing the Effectiveness and Security of the Use of Two Stentrievers Simultaneously Versus One Stentriever as a Primary Treatment in Acute Ischemic Stroke Patients.
Brief Title: Results of the Use of Two Stentrievers Simultaneosly Compared With One as a Primary Treatment in Acute Ischemic Stroke
Acronym: DIVERSO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPIC42
Record Dates: First submitted 2023-06-24; First posted 2023-07-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Thrombectomy; Arterial Occlusive Diseases
Keywords: Stroke; Double Stentriever; Thrombectomy
MeSH Terms: conditions — Stroke; Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patient & Outcomes adjudicator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double stentriever technique (Experimental): Patients treated with thrombectomy with a proximal balloon guiding catheter using two stentrievers simultaneously (one of 6 mm x 50 mm and another of 6 mm x 50 mm or 4 mm x 35 mm)
  Interventions: Device: Double stentriever
- Single stentriever technique (Active Comparator): Patients treated with thrombectomy with a proximal balloon guiding catheter using one stentriever (6 mm x 50 mm).
  Interventions: Device: Single stentriever

INTERVENTIONS:
Device: Double stentriever — Double stentriever technique
  Arms: Double stentriever technique
Device: Single stentriever — Single stentriever technique
  Arms: Single stentriever technique

SUMMARY:
Several studies have demonstrated that simultaneous treatment with two stentrievers (STs) as rescue treatment is very effective, with high recanalization rates even in this group of patients where other revascularization techniques have failed. There has been no observed increase in hemorrhagic complications. Recently, a prospective study has been published where treatment with two ST has been shown to be effective and safe if used as a first-choice treatment (not as rescue) with a successful recanalization rate (eTICI 2c/3) after the first pass of 69%. These results have been reinforced after the publication of a randomized study that confirms, in vitro, the superiority of using two ST over one.

DETAILED DESCRIPTION:
The use of a double stent retriever has been proposed as a safe and effective technique. The investigators hypothesized that the use of double stentriever primary could lead to higher first pass effect rates and better outcomes compared to single stentriever primary.

Our goal is to develop a research project to provide additional information on the potential benefits of the simultaneous double stent approach primarily in stroke patients receiving endovascular treatment.

A randomized study to compare the efficacy of double primary stentriever versus single primary stentriever.

ELIGIBILITY:
Inclusion Criteria:

* A new disabling focal neurological deficit compatible with acute cerebral ischemia.
* Any age. Informed consent obtained from the patient or representative.
* NIHSS score ≥ 6.
* Pre-existing functional clinical status less than or equal to 2 according to the mRS clinical scale.
* Maximum time of 24 hours from symptom onset to arterial puncture. • TICI 0-1 in the diagnosed TICA (terminal internal carotid artery) , MCA (middle cerebral artery), and BA( basilar artery confirmed by angioCT and angiography).
* ASPECTs score on baseline CT greater than or equal to 6.
* In cases where it is indicated, prior intravenous fibrinolysis will be administered according to the protocols of each center.

Exclusion Criteria:

* Those described in the usual protocols for mechanical thrombectomy of each hospital.
* Pre-existing functional clinical status greater than 2 according to the mRS clinical scale
* Patients with tandem lesions of dissection or arteriosclerotic origin located in the extracranial internal carotid artery.
* Initiation of treatment with a different technique than the one described.
* Inability to use a proximal balloon guide catheter.
* Use of aspiration catheter.
* Intracranial atherosclerotic plaque as the cause of occlusion.
* Advanced or terminal disease with a life expectancy of less than 6 months.
* Patient who is participating in another study that may affect this one.
* ASPECTS score less than or equal to 6 on baseline CT.
* Evidence of significant hemorrhage or mass effect with midline shift on baseline CT.
* Patients with occlusions in multiple vascular territories.
* Evidence of intracranial tumor (except for small meningiomas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
EFFECTIVENESS OBJECTIVE: Complete recanalization on first pass | 90 days
  Comparison of the complete recanalization rate in the first pass in the double stent group compared to the single stent group, defined as TICI greater than 2c on the Thrombolysis in Cerebral Infarction scale (eTICI scale).
SAFETY OBJECTIVE: Intracerebral hemorrhage. | 24 hours
  Rate of patients with symptomatic intracranial hemorrhage (neurological deterioration in National Institutes of Health Stroke Scale [NIHSS] >4) at 24h observed between both groups and, fundamentally, evaluated by CT.

SECONDARY OUTCOMES:
Intervention success. | During the procedure
  Rate of the ability to position both STs in the indicated location.
Complications related to the intervention. | During the procedure
  Evaluation of the rate of arterial perforation, angiographic extravasation of contrast, arterial dissection or arterial vasospasm.
Embolism in new territories. | During the procedure
  Rate of embolization to an artery not involved in the initially affected territory.
Number of passes with the devices. | During the procedure
  Evaluation of the number of passes with the devices during the procedure.
Procedure time. | During the procedure
  Time from arterial puncture to arterial recanalization, or if not achieved, until the end of the intervention.
Arterial Recanalization (eTICI scale) on first pass. | During the procedure
  evaluation of the rates of eTICI 3, eTICI 2c/3, eTICI e2b/3 on the Thrombolysis in Cerebral Infarction scale (e TICI scale); range 0-3, with highest score indicating complete recanalization.
Arterial recanalization at the end of the procedures. | During the procedure
  eTICI 3, eTICI e2c/3, eTICI e2b/3 at the end of the procedure on the Thrombolysis in Cerebral Infarction scale (e TICI scale); range 0-3, with highest score indicating complete recanalization.
Intracerebral hemorrhage. | 24 hours
  Rate of any type of intracranial hemorrhage on the 24-hour control computed tomography (CT) scan (subarachnoid hemorrhage and hemorrhage according to the classification used in the ECASS study).
Early neurological improvement. | 24 hours
  Rate of patients with a decrease of 10 points or more on the NIHSS scale or complete recovery during the first 24 hours. Improvement of Neurological status at 24 hours, determined by National Institutes of Health Stroke Scale [NIHSS score] range 0-42, with higher scores indicating greater stroke severity.
National Institutes of Health Stroke Scale (NIHSS) scale at 24 hours, on day 5, or at discharge. | 5 days
  Neurological status at 24 hours, at day 5 (+/- 12 hours) or discharge, determined by National Institutes of Health Stroke Scale [NIHSS score] range 0-42, with higher scores indicating greater stroke severity.
Modified Rankin Scale (mRS) scale at 90 days. | 90 days
  Modified Rankin Scale (mRS; range 0 [no symptoms] to 6 [death] for the evaluation of neurological functional disability score at 90 days
Mortality rate. | 90 days
  90-day mortality rate.

CONTACTS AND LOCATIONS:
Locations (4):
- Alfried Krupp Hospital Ruettenscheid, Essen, Germany
- Spain (3):
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vega P, Murias E, Jimenez JM, Chaviano J, Rodriguez J, Calleja S, Delgado M, Benavente L, Castanon M, Puig J, Cigarran H, Arias F, Chapot R. First-line Double Stentriever Thrombectomy for M1/TICA Occlusions : Initial Experiences. Clin Neuroradiol. 2022 Dec;32(4):971-977. doi: 10.1007/s00062-022-01161-2. Epub 2022 Apr 13. PMID 35416489
- [Background] Li J, Tiberi R, Canals P, Vargas D, Castano O, Molina M, Tomasello A, Ribo M. Double stent-retriever as the first-line approach in mechanical thrombectomy: a randomized in vitro evaluation. J Neurointerv Surg. 2023 Dec;15(12):1224-1228. doi: 10.1136/jnis-2022-019887. Epub 2023 Jan 10. PMID 36627194
- [Background] Okada H, Matsuda Y, Chung J, Crowley RW, Lopes DK. Utility of a Y-configured stentriever technique as a rescue method of thrombectomy for an intractable rooted thrombus located on the middle cerebral artery bifurcation: technical note. Neurosurg Focus. 2017 Apr;42(4):E17. doi: 10.3171/2017.1.FOCUS16511. PMID 28366064
- [Background] Cabral LS, Mont'Alverne F, Silva HC, Passos Filho PE, Magalhaes PSC, Bianchin MM, Nogueira RG. Device size selection can enhance Y-stentrieving efficacy and safety as a rescue strategy in stroke thrombectomy. J Neurointerv Surg. 2022 Jun;14(6):558-563. doi: 10.1136/neurintsurg-2021-017751. Epub 2021 Jul 7. PMID 34233944
- [Background] Li Z, Liu P, Zhang L, Zhang Y, Fang Y, Xing P, Huang Q, Yang P, Liu J. Y-Stent Rescue Technique for Failed Thrombectomy in Patients With Large Vessel Occlusion: A Case Series and Pooled Analysis. Front Neurol. 2020 Aug 27;11:924. doi: 10.3389/fneur.2020.00924. eCollection 2020. PMID 32973671